CLINICAL TRIAL: NCT03917550
Title: RECOVERY: An Internet-delivered Transdiagnostic Cognitive Behavior Therapy in Romania
Brief Title: RECOVERY: A Transdiagnostic Intervention for Anxiety and Depression
Acronym: RECOVERY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUT - RECOVERY
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Depression; Dysthymic Disorder; Panic Disorder; Social Phobia; Generalized Anxiety Disorder; Specific Phobia
Keywords: Transdiagnostic; Cognitive behavioural therapy (CBT); Depression; Anxiety
MeSH Terms: conditions — Depression; Dysthymic Disorder; Panic Disorder; Phobia, Social; Generalized Anxiety Disorder; Phobia, Specific; Anxiety Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Folow-up interviews will be carried out by a different team of assessors (blinded to the treatment condition)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery (Transdiagnostic & self) (Experimental): A longitudinal study conducted before has shown that self-compassion, unconditional self-acceptance, self-esteem and self concept clarity could be considered risk factors for the severity of the clinical symptoms in anxiety and depression. This is the main reason why this arm consists of the Transdiagnostic intervention program for emotional disorders plus a number of intervention techniques targeting the self-concepts mentioned before. The intervention, based on the Cognitive Behavioral Therapy (CBT) principles, is designed to encourage participants to confront and experience uncomfortable emotions, and use adaptive coping mechanisms. Moreover, additional intervention techniques targeting self-concepts will be used to improve participants' self.
  Interventions: Behavioral: Recovery (Transdiagnostic & self)
- Transdiagnostic (Active Comparator): This arm represents the Transdiagnostic intervention program for emotional disorders. The intervention, based on the Cognitive Behavioral Therapy (CBT) principles, is designed to encourage participants to confront and experience uncomfortable emotions, and use adaptive coping mechanisms.
  Interventions: Behavioral: Transdiagnostic

INTERVENTIONS:
Behavioral: Recovery (Transdiagnostic & self) — This transdiagnostic program is based on the general Cognitive Behavioral Therapy (CBT) principles and targets core higher order factors such as negative affectivity and emotion dysregulation, using common intervention techniques applicable across disorders. The program was designed to directly address the aversive emotional experiences often reported by clients, hoping to reverse participants' maladaptive thinking style and dysfunctional behaviors. In addition, specific intervention designed to improve self-compassion, unconditional self-acceptance, self-esteem and self concept clarity were added.
  Arms: Recovery (Transdiagnostic & self)
Behavioral: Transdiagnostic — This transdiagnostic program is based on the general Cognitive Behavioral Therapy (CBT) principles and targets core higher order factors such as negative affectivity and emotion dysregulation, using common intervention techniques applicable across disorders. The program was designed to directly address the aversive emotional experiences often reported by clients, hoping to reverse participants' maladaptive thinking style and dysfunctional behaviors.
  Arms: Transdiagnostic

SUMMARY:
To investigate the efficacy and acceptability of a guided internet delivered transdiagnostic intervention, targeting mild to moderate clinical symptoms of anxiety and depression and emphasizing the changes taking place at the level of the structures of the self.

DETAILED DESCRIPTION:
The effectiveness of a Transdiagnostic Cognitive-Behavioral Treatment will be compared with an improved version of it, in which new intervention techniques were added, pointing out the importance of improving some self-concept dimensions in reducing symptoms of anxiety and depression. In order to prove this, the study design will include two active intervention groups; a standard transdiagnostic intervention protocol will be delivered to one group and an improved version of the same transdiagnostic protocol will be delivered to the other group. The new added techniques targets some self-concepts, namely self-compassion, unconditional self-acceptance and self-esteem. The main goal of the study is to concurrently test effectiveness of these two transdiagnostic approaches in reducing symptoms of anxiety and depression and improving the above-mentioned self-concepts. This non-inferiority trial has the power to detect an effect size larger than Cohen's d = .40 (including 20% attrition at post-test and 6 month follow-up)

ELIGIBILITY:
Inclusion Criteria:

1. be fluent in Romanian,
2. be at least 18 years of age,
3. have at least a clinical diagnosis of major depressive disorder/dysthymia, and/or generalized anxiety disorder, and/or social anxiety disorder, panic anxiety disorder and/or Agoraphobia, specific phobia or any combination of these conditions on Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders 5 (SCID-I 5)

Exclusion Criteria:

1. suicidal plans,
2. changes in the dosage if psychotropic medication during the last month (if present),
3. have bipolar disorder or psychosis (according to medication status),
4. have an alcohol/substance abuse and/or dependence disorder,
5. currently take part in other psychological treatment,
6. obvious obstacle to participation (i.e., no current Internet access, long travel plans during the treatment period etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-03-27 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ9) | Absolute values (average score) of PHQ9 at 10 weeks (post-intervention)
  The Patient Health Questionnaire 9 (PHQ9) was designed to measure participant's level of depression. The scale is unidimensional and the total score ranges from 0 to 27. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
Generalized Anxiety Disorder 7 (GAD7) | Absolute values (average score) of GAD7 at 10 weeks (post-intervention)
  Generalized Anxiety Disorder 7 (GAD7) was designed to measure participant's level of generalized anxiety or worry. The scale is unidimensional and the total score ranges from 0 to 21. Low scores are associated with low levels of worry, while high scores are associated with high levels of worry.
Social Phobia Inventory (SPIN) | Absolute values (average score) of SPIN at 10 weeks (post-intervention)
  The SPIN was designed to measure participant's level of social phobia. The scale is unidimensional and the total score ranges from 0 to 68. Low scores are associated with low levels of social phobia, while high scores are associated with high levels of social phobia.
Panic Disorder Severity Scale-Self Report (PDSS-SR) | Absolute values (average score) of PDSS-SR at 10 weeks (post-intervention)
  The PDSS-SR was designed to measure participant's level of panic. The scale is unidimensional and the total score rages from 0 to 28. Low scores are associated with low levels of panic, while high scores are associated with high levels of panic.

SECONDARY OUTCOMES:
Work and Social Adjustment Scale (WSAS) | Absolute values (average score) of WSAS at 10 weeks (post-intervention)
  Work and Social Adjustment Scale (WSAS) was designed to measure symptom interference. The scale is unidimensional and the total score ranges from 0 to 40. Low scores are associated with higher levels of functioning (less interference of clinical symptoms) while high scores are associated with lower levels of functioning (or high interference of clinical symptoms).
Beck Depression Inventory-II (BDI-II) | Absolute values (average score) of BDI-II at 10 weeks (post-intervention)
  The Beck Depression Inventory-II (BDI-II) was designed to measure participant's level of depression. The scale is unidimensional and the total score ranges from 0 to 63. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
Penn State Worry Questionnaire (PSWQ) | Absolute values (average score) of PSWQ at 10 weeks (post-intervention)
  The PSWQ was designed to measure participant's level of generalized anxiety or worry. The scale is unidimensional and the total score ranges from 16 to 80. Low scores are associated with low levels of worry, while high scores are associated with high levels of worry.
Anxiety Sensitivity Index 16 (ASI16) | Absolute values (average score) of ASI at 10 weeks (post-intervention)
  The ASI was designed to measure participant's level of anxiety sensitivity. The scale is unidimensional and the total score rages from 0 to 64. Low scores are associated with low levels of anxiety sensitivity, while high scores are associated with high levels of anxiety sensitivity.
Self-Concept Clarity Scale (SCCS) | Absolute values (average score) of SCCS at 10 weeks (post-intervention)
  SCCS was designed to measure participant's level of their Self-Concept Clarity. The scale is unidimensional and the total score rages from 12 to 60. Low scores are associated with low levels of Self-Clarity, while high scores are associated with high levels of Self-Clarity.
New General Self-Efficacy Scale (NGSE) | Absolute values (average score) of NGSE at 10 weeks (post-intervention)
  NGSE was designed to measure participant's level of Self-Efficacy. The scale is unidimensional and the total score rages from 8 to 40. Low scores are associated with low levels of Self-Efficacy, while high scores are associated with high levels of Self-Efficacy.
Unconditional Self-Acceptance Questionnaire (USAQ) | Absolute values (average score) of USAQ at 10 weeks (post-intervention)
  USAQ was designed to measure participant's level of unconditional Self-Acceptance. The scale is unidimensional and the total score rages from 20 to 140. Low scores are associated with low levels of unconditional Self-Acceptance, while high scores are associated with high levels of unconditional Self-Acceptance.
Overall Anxiety Severity and Impairment Scale (OASIS) | Absolute values (average score) of OASIS at 10 weeks (post-intervention)
  The OASIS was designed to measure participant's level of overall anxiety level. The scale is unidimensional and the total score rages from 0 to 20. Low scores are associated with low levels of anxiety, while high scores are associated with high levels of anxiety.
Overall Depression Severity and Impairment Scale (ODSIS) | Absolute values (average score) of ODSIS at 10 weeks (post-intervention)
  The ODSIS was designed to measure participant's level of overall depression level. The scale is unidimensional and the total score rages from 0 to 20. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
Rosenberg Self-Esteem Scale (RSES) | Absolute values (average score) of RSES at 10 weeks (post-intervention)
  Rosenberg Self-Esteem Scale was designed to measure participant's level of Self-Esteem. The scale is unidimensional and the total score rages from 10 to 40. Low scores are associated with low levels of Self-Esteem, while high scores are associated with high levels of Self-Esteem.
Self-Compassion Scale (SCS) | Absolute values (average score) of SCS at 10 weeks (post-intervention)
  SCS was designed to measure participant's level of their Self-Compassion. The scale is multidimensional and the total score rages from 26 to 130. Low scores are associated with low levels of Self-Compassion, while high scores are associated with high levels of Self-Compassion.
Minnesota Multiphasic Personality Inventory 2 Neagtive Treatment Indicator Scale (MMPI2TRT) | Absolute values (average score) of MMPI2TRT at 10 weeks (post-intervention)
  MMPI2TRT was designed to measure participants negative attitudes toward doctors/mental health professionals and unwilling to discuss personal problems. The scale is unidimensional and the total score rages from 0 to 26. Low scores are associated positive attitudes towards doctors and willingness to discuss problems while high scores are associated with negative attitudes toward doctors and unwilling to discuss personal problems.
Personality Clinical Form - Neagtive TReaTment Indicator Scale (PCFTRT) | Absolute values (average score) of PCFTRT at 10 weeks (post-intervention)
  PCFTRT is a new subscale designed to assess participants negative attitudes toward mental health professionals and unwilling to discuss personal problems. The subscale is unidimensional and the total score rages from 0 to 24. Low scores are associated positive attitudes towards doctors and willingness to discuss problems while high scores are associated with negative attitudes toward doctors and unwilling to discuss personal problems.

CONTACTS AND LOCATIONS:
Overall Officials: Andreea Isbasoiu, PhD student, Study Director — West University of Timisoara
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No
Data will be process only at the group level. No individual data will be shared to third parties.

REFERENCES:
- [Derived] Isbasoiu AB, Tulbure BT, Rusu A, Sava FA. Can We Boost Treatment Adherence to an Online Transdiagnostic Intervention by Adding Self-Enhancement Strategies? Results From a Randomized Controlled Non-inferiority Trial. Front Psychol. 2021 Dec 2;12:752249. doi: 10.3389/fpsyg.2021.752249. eCollection 2021. PMID 34925157
- See also: Project official website — https://www.e-cbt.ro/program/recovery